CLINICAL TRIAL: NCT01686945
Title: Investigation on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of a Long-acting GLP-1 Analogue in Healthy Male Subjects and Male Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-3991; 2012-000361-20 (EudraCT Number); U1111-1127-4408 (Other: WHO)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy - 20 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Healthy - 40 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Healthy - 60 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- T2D - 20/40/60 mg (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Start doses of 5 mg and 10 mg with end dose of 20 mg. For oral administration.
  Arms: Healthy - 20 mg
Drug: semaglutide — Start doses of 5 mg and 10 mg with end doses of either 20 mg or 40 mg. For oral administration.
  Arms: Healthy - 40 mg
Drug: semaglutide — Start doses of 5 mg and 10 mg with end doses of either 20 mg, 40 mg or 60 mg. For oral administration.
  Arms: Healthy - 60 mg; T2D - 20/40/60 mg
Drug: placebo — Placebo semaglutide. For oral administration.
Drug: placebo — Placebo semaglutide with carrier. For oral administration.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body), and pharmacodynamics (the effect of the investigated drug on the body) of multiple doses of a long-acting GLP-1 analogue (oral semaglutide) and a carrier in healthy male subjects and male subjects with type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Male subject, who is considered to be generally healthy, based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and laboratory safety tests performed during the screening visit, as judged by the investigator. This also applies to subjects with T2D, except for the underlying diabetes with or without associated hyperlipidaemia and/or hypertension
* Body mass index (BMI): a) Healthy subjects: above or equal to 20 and below 30 kg/m^2. b) Subjects with T2D: BMI above or equal to 20 and below or equal to 37 kg/m^2
* Glycosylated haemoglobin (HbA1c): a) Healthy subjects: below 6.0%. b) Subjects with T2D: between 6.5 and 9.0% (both inclusive)
* Additional inclusion criterion only for subjects with T2D: Male subjects with T2D (diagnosed within the past 10 years) treated with diet and exercise and/or who have been on stable doses of metformin for at least 12 weeks prior to Visit 3 (Day -1 or 0) and for whom no changes in treatment are planned for the trial period

Exclusion Criteria:

* History of, or presence of, cancer, diabetes (only for healthy subjects) or any clinically significant cardiovascular (only for healthy subjects), respiratory, metabolic, renal, hepatic, gastro-intestinal (GI), endocrinological (except diabetes in subjects with T2D), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Blood pressure in supine position at the screening examination above: a) 140 mmHg systolic and/or above 90 mmHg diastolic for healthy subjects. b) 160 mmHg systolic and/or above 95 mmHg diastolic for subjects with T2D
* Use of prescription or non-prescription medicinal products (except routine vitamins) within three weeks preceding the dosing. Occasional use of paracetamol or acetylsalicylic acid is permitted. a. For subjects with T2D: Any other current diabetes treatment apart from metformin (e.g. treatment with incretin mimetics, Dipeptidyl Peptidase-IV (DPP-IV) inhibitors, insulin secretagogues, insulin or thiazolidinediones (TZDs)). Use of blood lipidregulating agents, as well as blood pressure regulating, and thrombo-embolic agents is allowed
* Exclusion criteria only for subjects with T2D:
* Proliferative retinopathy or maculopathy requiring acute treatment as determined by funduscopy/fundus photography and judged by the investigator. If subject presents a medical certificate for funduscopy/fundus photography performed within last 3 months this can substitute the funduscopy/fundus photography at screening
* Nephropathy stages 3 to 5, i.e. estimated glomerular filtration rate (eGFR) below 60. The eGFRshould be determined using the Modification of Diet in Renal Disease 4-variable method encompassing creatinine, age, gender, and race
* Diabetic peripheral neuropathy using the 10 g Semmes-Weinstein monofilament examination at the great toe or plantar aspect of the fifth metatarsal
* Clinically significant active cardiovascular disease including history of myocardial infarction and/or heart failure (New York Heart Association (NYHA) class III and IV1) at the discretion of the investigator

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2013-04-08 (Actual); Study Completion 2013-04-08 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) recorded | From the time of first dosing and until completion of the post treatment follow-up visits (Day 90 to 104)

SECONDARY OUTCOMES:
Area under the plasma concentration curve over the dosing interval (0-24 hours) | After the last 3 daily doses for semaglutide and carrier
Change from baseline in fasting plasma glucose (FPG) | Week 0, week 10 (Day 69)
Change from baseline in C-peptide | Week 0, week 10 (Day 69)
Change from baseline in insulin | Week 0, week 10 (Day 69)
Change from baseline in glucagon | Week 0, week 10 (Day 69)
Change from baseline in glycosylated haemoglobin type A1c (HbA1c) | Week 0, week 10 (Day 69)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] Seco A, Aparicio S, Gonzalez-Camejo J, Jimenez-Benitez A, Mateo O, Mora JF, Noriega-Hevia G, Sanchis-Perucho P, Serna-Garcia R, Zamorano-Lopez N, Gimenez JB, Ruiz-Martinez A, Aguado D, Barat R, Borras L, Bouzas A, Marti N, Paches M, Ribes J, Robles A, Ruano MV, Serralta J, Ferrer J. Resource recovery from sulphate-rich sewage through an innovative anaerobic-based water resource recovery facility (WRRF). Water Sci Technol. 2018 Dec;78(9):1925-1936. doi: 10.2166/wst.2018.492. PMID 30566096
- [Derived] Granhall C, Donsmark M, Blicher TM, Golor G, Sondergaard FL, Thomsen M, Baekdal TA. Safety and Pharmacokinetics of Single and Multiple Ascending Doses of the Novel Oral Human GLP-1 Analogue, Oral Semaglutide, in Healthy Subjects and Subjects with Type 2 Diabetes. Clin Pharmacokinet. 2019 Jun;58(6):781-791. doi: 10.1007/s40262-018-0728-4. PMID 30565096
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com